CLINICAL TRIAL: NCT02587338
Title: Verbesserung Kognitiver Fähigkeiten im Alter
Brief Title: Cognitive Ability Training in Seniors
Acronym: CATS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Wuerzburg22/15
Record Dates: First submitted 2015-06-16; First posted 2015-10-27 (Estimated); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Mild Cognitive Impairment
Keywords: Subjective Memory Impairment; tDCS; NIRS; Cognitive Training; Working Memory
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Verum tDCS (Experimental): Left frontal anodal stimulation, supraorbital right cathodal stimulation
  Interventions: Device: Verum tDCS
- Sham tDCS (Experimental): sham stimulation, same electrode positions
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Verum tDCS — Neuropsychological (Working memory) training for 30 minutes, 6 sessions tDCS during training with 2000 microampere left anodal, right cathodal
  Arms: Verum tDCS
Device: Sham tDCS — Neuropsychological (Working memory) training for 30 minutes, 6 sessions tDCS during training with 0 microampere
  Arms: Sham tDCS

SUMMARY:
This study investigates the beneficial effects of prefrontal brain stimulation (with transcranial direct current stimulation [tDCS]) during working memory training in seniors with subjective memory impairments.The placebo-controlled double blinded study includes 50 elderly probands which were randomized into verum or sham tDCS.

ELIGIBILITY:
Inclusion Criteria:

* native german speaker
* between 60-70 years old
* subjective memory impairment

Exclusion Criteria:

* psychiatric, neurological diseases
* uncorrected hearing or vision deficits
* actual psychopharmaco intake
* metal parts in the head
* medical electronical implants

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin J. Herrmann, PD Dr, Principal Investigator — University of Würzburg
Locations (1):
- University hospital, Würzburg, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Verum tDCS: Left frontal anodal stimulation, supraorbital right cathodal stimulation
  Verum tDCS: Neuropsychological (Working memory) training for 30 minutes, 6 sessions tDCS during training with 2000 microampere left anadal, right cathodal
Period: Overall Study
Arm/Group | Verum tDCS | Sham tDCS
Started | 20 | 18
Completed | 20 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Verum tDCS | Sham tDCS | Total
Number analyzed (Participants) | 20 | 18 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (3.0) | 64.2 (2.5) | 64.2 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 27
  Male | 5 | 6 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 20 | 18 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 20 | 18 | 38

OUTCOME MEASURES:

1. Primary Outcome: Neuropsychological Performance in Neuropsychological Test: Verbal Learning Memory Test (VLMT)
Description: The Investigators are measuring cognitive performance for different executive functions, here the score (percentile of the norm values) of the test verbal learning memory test (VLMT), parameter immediate recall post treatment is reported. Rage from 0 to 100 %. Higher values indicate higher performance.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Verum tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 18
score on a scale | 57.2 (9.4) | 57.2 (5.1)
Statistical Analysis 1: Comparison: Verum tDCS vs Sham tDCS; Test type: Superiority; p = 0.74, ANOVA

2. Secondary Outcome: Brain Activation Measured With Near-infrared Spectroscopy (NIRS) During the Semantic Condition of the Verbal Fluency Task (VFT)
Description: NIRS is a brain imaging method, with the parameters of oxy (OxyHB) and deoxy (deoxyHB) hemoglobin. Activation is reflected by increase of OxyHB and decrease DeoxyHB. Differences from pre- to post-measurement for OxyHB are reported in a region of interest analysis of the dorsolateral prefrontal cortex.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Unit of Measure: Δ mol/L
Arm/Group | Verum tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 18
Unit of Measure: Δ mol/L | -12.43 (13.37) | -3.68 (14.66)
Statistical Analysis 1: Comparison: Verum tDCS vs Sham tDCS; Test type: Superiority; p = 0.062, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Verum tDCS | Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/18
Other Adverse Events (participants affected / at risk) | 0/20 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes